CLINICAL TRIAL: NCT02152150
Title: Efficacy of Iron Bio-fortified Pearl Millet in Improving the Iron Status of Adolescents in India
Brief Title: Feeding Trial of Bio-fortified Pearl Millet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: SNDT Women's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB #: 1107002349
Record Dates: First submitted 2014-05-13; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Iron Deficiency and Anemia
Keywords: iron; anemia; bio-fortification; children; India
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron bio-fortified pearl millet (Experimental): Pearl millet variety ICTP8203-Fe (82 mg/kg iron content)
  Interventions: Other: Iron bio-fortified pearl millet
- Control pearl millet (Active Comparator): Conventional pearl millet: variety DG9444 (22 mg/kg iron content) and JKBH778 (52 mg/kg iron content)
  Interventions: Other: Control pearl millet

INTERVENTIONS:
Other: Iron bio-fortified pearl millet — Pearl millet variety ICTP8203-Fe (82 mg/kg iron content) prepared as a traditional flatbread (bhakri)
  Arms: Iron bio-fortified pearl millet
Other: Control pearl millet — Conventional pearl millet: variety DG9444 (22 mg/kg iron content) and JKBH778 (52 mg/kg iron content), prepared as a traditional flatbread (bhakri)
  Arms: Control pearl millet

SUMMARY:
The objective of this study was to evaluate the efficacy of iron bio-fortified pearl millet in improving iron status in adolescents in India.

DETAILED DESCRIPTION:
An estimated 1.6 billion people worldwide are anemic, and iron deficiency (ID) is the leading cause of anemia. Its prevalence is highest in resource-limited settings, and among children and women of reproductive age. Even mild ID can adversely impact cognitive performance, behavior, and physical growth of children, and physical work and cognitive performance in adults.

Interventions to target micronutrient malnutrition such as dietary diversification, micronutrient supplementation, and food fortification have reduced ID, but have not been universally successful. Biofortification, the process of increasing the concentration and bioavailability of essential nutrients in staple crops by traditional plant breeding, is a sustainable and cost-effective approach to combat micronutrient deficiencies. Other forms of bio-fortification (agronomic management and genetic modification) are also feasible. Rice, maize, wheat, pearl millet, sweet potato, beans, and cassava have been the main target crops of bio-fortification.

Pearl millet (PM) is a primary staple food in India, particularly in the states of Rajasthan, Gujarat and Maharashtra. The high pearl millet consumption and availability of a recently released pearl millet variety (ICTP 8203-Fe) with significantly greater iron content provided an opportunity to evaluate its efficacy on improving iron status in human populations. We hypothesized that daily consumption of iron bio-fortified pearl millet (Fe-PM) would improve iron status in six months. We conducted a randomized efficacy trial of iron bio-fortified pearl millet in improving iron status in adolescents in Maharashtra, India.

The aims of this study are:

* To determine if the iron status of adolescent boys and girls in rural Maharashtra is improved by consuming high-iron bio-fortified PM
* To determine if adolescents in rural Maharashtra consuming high-iron bio-fortified PM exhibit higher physical performance and energetic work efficiency compared to adolescent boys and girls consuming low-iron pearl millet.
* To determine if adolescents in rural Maharashtra consuming high-iron bio-fortified PM exhibit higher cognitive and perceptual functioning, as well as differences in patterns of cortical activation' when compared to children consuming low-iron pearl millet.

The principal hypotheses to be tested are that in an intervention study using iron bio-fortified PM with the highest possible levels of iron content in comparison to a low-iron control:

* Iron bio-fortified PM consumed as a dietary iron intervention will improve the iron status of iron deficient adolescents
* Iron bio-fortified PM consumed as a dietary iron intervention will improve the physical performance of iron deficient adolescents
* Iron bio-fortified PM as an iron intervention will improve the cognitive and perceptual functioning of iron deficient adolescents

The long-term goal of this study is to show that iron bio-fortification of PM is an efficacious and potentially effective strategy for addressing iron deficiency in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Participants are individuals aged 12 to 16 years
* Attending boarding schools in Ahmednagar district, Maharashtra, India

Exclusion Criteria:

* Severe anemia (Hemoglobin<8.5g/dL)
* Taking iron supplements or medications that could interfere with iron absorption
* Chronic illnesses

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in iron status | 6 months
  Hemoglobin, serum ferritin, serum transferrin receptor, body iron

SECONDARY OUTCOMES:
Differences in cognitive function | 6 months
  Five tests of perceptual and cognitive performance: i) the simple reaction time task; ii) the go-nogo task; iii) the attentional network task; iv) the composite face task; and v) the cued recognition memory task.
  Approximately 1/2 of participants performed these tasks with concurrent recording of electroencephelography (EEG).
Differences in physical performance | 6 months
  i) estimation of maximal oxygen consumption, ii) determination of energy expenditure and work efficiency at modest levels of exertion, and iii) determination of time spent at 3 levels of physical exertion while performing normal daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jere D. Haas, Ph.D., Principal Investigator — Cornell University; Shobha Udipi, Ph.D., Principal Investigator — SNDT Women's University
Locations (1):
- S.N.D.T. Women's University, Mumbai, India

REFERENCES:
- [Derived] Wenger MJ, Murray Kolb LE, Scott SP, Boy E, Haas JD. Modeling relationships between iron status, behavior, and brain electrophysiology: evidence from a randomized study involving a biofortified grain in Indian adolescents. BMC Public Health. 2022 Jul 6;22(1):1299. doi: 10.1186/s12889-022-13612-z. PMID 35794587
- [Derived] Scott SP, Murray-Kolb LE, Wenger MJ, Udipi SA, Ghugre PS, Boy E, Haas JD. Cognitive Performance in Indian School-Going Adolescents Is Positively Affected by Consumption of Iron-Biofortified Pearl Millet: A 6-Month Randomized Controlled Efficacy Trial. J Nutr. 2018 Sep 1;148(9):1462-1471. doi: 10.1093/jn/nxy113. PMID 30016516
- [Derived] Finkelstein JL, Mehta S, Udipi SA, Ghugre PS, Luna SV, Wenger MJ, Murray-Kolb LE, Przybyszewski EM, Haas JD. A Randomized Trial of Iron-Biofortified Pearl Millet in School Children in India. J Nutr. 2015 Jul;145(7):1576-81. doi: 10.3945/jn.114.208009. Epub 2015 May 6. PMID 25948782